CLINICAL TRIAL: NCT01700621
Title: Non-interference and Safety of Concomitant Administration of Measles-rubella and Rotavirus Vaccines at 9 Months of Age in Rural Bangladesh
Brief Title: Coadministration of Measles-rubella and Rotavirus Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS677
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Measles Antibody Seroconversion; Rubella Antibody Seroconversion; Rotavirus Geometric Mean Titer (GMT); Rotavirus Immunoglobulin A (IgA) Seropositivity
Keywords: rotavirus
MeSH Terms: interventions — RIX4414 vaccine; Rotavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- measles-rubella and rotavirus vaccines (Experimental): receive one 0.5 ml subcutaneous dose of live attenuated measles-rubella vaccine and one 1.0 ml dose of oral Rotarix vaccine at 9 months of age
  Interventions: Biological: Rotarix vaccine; Biological: measles-rubella vaccine
- measles-rubella vaccine (Active Comparator): receive one 0.5 ml subcutaneous dose of live attenuated measles-rubella vaccine at 9 months of age
  Interventions: Biological: measles-rubella vaccine

INTERVENTIONS:
Biological: Rotarix vaccine — one 1.0 ml dose of oral rotavirus vaccine at 9 months of age
  Other Names: rotavirus vaccine
  Arms: measles-rubella and rotavirus vaccines
Biological: measles-rubella vaccine — one 0.5 ml subcutaneous dose of live attenuated measles-rubella vaccine
  Other Names: Measles-Rubella Virus Vaccine Live US Pharmacopeia (USP)

SUMMARY:
The investigators aim to establish the non-inferiority of concomitant administration of measles-rubella and rotavirus vaccines to measles-rubella vaccine given alone in terms of measles seroconversion rates. The primary study hypothesis is the measles seroconversion rate as defined by the percentage of children seroconverting to measles with a measles serum antibody concentration of >=1:120 at 8 weeks post vaccination after the concomitant administration of measles-rubella and rotavirus vaccines is non-inferior to that obtained when measles-rubella vaccine is given alone in children 9 months of age who have received a primary rotavirus vaccine series with the first dose between 6 and 10 weeks and the second at least 4 weeks later and are seronegative for measles antibody in the pre-vaccination sample.

ELIGIBILITY:
Inclusion Criteria:

* Child 9 months of age eligible for measles-rubella vaccination
* documented evidence of a primary rotavirus vaccine series with first dose between 6 and 10 weeks of age and second dose at least 4 weeks after first dose
* healthy infants free of chronic or serious medical condition as determined by history and physical examination at time of study enrollment
* parents/guardians of each participant are able to understand and follow study procedures and agree to participate in study by providing signed informed consent

Exclusion Criteria:

* hypersensitivity to any component of measles-rubella or Rotarix vaccine which would preclude administration of the vaccine
* history of intussusception, intestinal malformations, or abdominal surgery
* known history of measles and/or rubella disease
* history of previous receipt of measles and/or rubella vaccine
* use of any immunosuppressive drugs or immunoglobulin and/or blood products since birth or anticipated during study period
* current enrolment in any other intervention trial or use of any investigational drug or vaccine throughout the study period
* any participant who reports planning to leave the study area before the completion of the study
* acute diarrhea (defined as ≥3 loose stools within a 24-hour period) or vomiting (defined as projectile vomiting or any vomiting at the discretion of the clinician) at the time of enrollment or within the last 24 hours
* acute febrile illness (defined as a temperature of ≥38°C) at the time of enrollment.

Ages: 9 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 482 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K Zaman, PhD, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Zaman K, Fleming JA, Victor JC, Yunus M, Bari TI, Azim T, Rahman M, Mowla SM, Bellini WJ, McNeal M, Icenogle JP, Lopman B, Parashar U, Cortese MM, Steele AD, Neuzil KM. Noninterference of Rotavirus Vaccine With Measles-Rubella Vaccine at 9 Months of Age and Improvements in Antirotavirus Immunity: A Randomized Trial. J Infect Dis. 2016 Jun 1;213(11):1686-93. doi: 10.1093/infdis/jiw024. Epub 2016 Jan 27. PMID 26823338

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study population was drawn from participants living in the International Center for Diarrheal Disease Research, Bangladesh (icddr,b) service area of Matlab, Bangladesh.
Pre-assignment Details: Recruitment concurrently conducted at a number of health sites in the study area, which resulted in two additional infants being enrolled but subsequently not vaccinated with withdrawn from the study.
Period: Received Study Vaccines
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Started | 240 | 240
Completed | 240 | 240
Not Completed | 0 | 0
Period: Analyzed for Immunogenicity
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Started | 240 | 240
Completed | 227 | 233
Not Completed | 13 | 7
Not completed — Lost to Follow-up | 7 | 4
Not completed — Protocol Violation | 5 | 1
Not completed — Baseline measles measure high | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine | Total
Number analyzed (Participants) | 240 | 240 | 480
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.38 (0.252) | 9.39 (0.254) | 9.38 (0.253)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 123 | 233
  Male | 130 | 117 | 247
Currently breastfed [Count of Participants; unit: Participants]
  Yes | 236 | 238 | 474
  No | 4 | 2 | 6
Length [Mean (Standard Deviation); unit: cm] | 69.56 (2.488) | 69.81 (2.786) | 69.68 (2.642)
Weight [Mean (Standard Deviation); unit: kilograms] | 8.01 (1.101) | 7.97 (0.933) | 7.99 (1.047)
Mother's age [Mean (Standard Deviation); unit: years] | 27.1 (5.84) | 26.7 (5.90) | 26.9 (5.87)

OUTCOME MEASURES:

1. Primary Outcome: Percentage/Number of Subjects With Seroprotection for Measles Virus Serum Neutralization Antibodies
Description: Detected by plaque reduction neutralization test (PRNT).
  Seroprotection defined as measles serum antibody concentration >=1:120 8 weeks post vaccination. Assays were standardized using WHO Second International Standard for measles antibody containing 5000 mIU/ml, which enables the 50% neutralizing antibody end-point dose (titer, ND50) of test samples to be transformed to antibody concentrations in terms of mIU/ml. The analytical cut-off value in this assay was ND50 < 1/8; this was the lowest dilution at which sera were tested.
Time Frame: 8 weeks post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 227 | 233
Participants
  Seroprotection | 171 | 173
  No seroprotection | 56 | 60
Statistical Analysis 1: Comparison: Measles-rubella and Rotavirus Vaccines vs Measles-rubella Vaccine; Test type: Non-Inferiority — A noninferiority margin of -10% was chosen as the maximal absolute reduction in proportion seroprotection allowed in the concomitant measles-rubella and rotavirus vaccine group as compared to the measles-rubella vaccine alone group; Seroconversion proportion difference = 1.1, 95% CI 2-sided [-6.9 to 9.0]

2. Primary Outcome: Percentage/Number of Subjects With Seroprotection for Anti-measles Virus Immunoglobulin G (IgG)
Description: Used commercially available indirect enzyme-linked IgG immunoassays (EIAs; Wampole Laboratories, Princeton, New Jersey). An index standard ratio (ISR) of ≥1.10 on both runs of the respective assay was considered evidence of seropositivity for measles virus. All measles virus and rubella virus assays were performed at the National Measles and Rubella Reference Laboratories, Measles, Mumps, Rubella, and Herpesviruses Branch, Division of Viral Diseases, Centers for Disease Control and Prevention (Atlanta, Georgia).
Time Frame: 8 weeks post vaccination
Population: All children meeting inclusion/exclusion criteria with a valid sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 227 | 232
Participants
  Seroprotection | 219 | 227
  No seroprotection | 8 | 5

3. Secondary Outcome: Percentage/Number of Subjects With Seroconversion for Anti-rubella Virus Immunoglobulin G (IgG)
Description: Used commercially available indirect enzyme-linked IgG immunoassays (EIAs; Wampole Laboratories, Princeton, New Jersey). An index standard ratio (ISR) of ≥1.10 on both runs of the respective assay was considered evidence of seropositivity for rubella virus. An ISR of at least 1.10 represents 10 IU/mL of rubella virus antibody, consistent with a protective level.All measles virus and rubella virus assays were performed at the National Measles and Rubella Reference Laboratories, Measles, Mumps, Rubella, and Herpesviruses Branch, Division of Viral Diseases, Centers for Disease Control and Prevention (Atlanta, Georgia).
Time Frame: 8 weeks post vaccination
Population: All children meeting inclusion and exclusion criteria with valid samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 228 | 234
Participants
  Seroprotection | 228 | 233
  No seroprotection | 0 | 1

4. Secondary Outcome: Geometric Mean Concentration (GMC) for Anti-rubella Virus Immunoglobulin G (IgG)
Description: as for outcome 3
Time Frame: 8 weeks post vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 228 | 234
IU/mL | 191.9 [174.8 to 210.7] | 177.8 [161.8 to 195.4]

5. Secondary Outcome: Percentage/Number of Subjects Seropositive for Anti-rotavirus Immunoglobulin A (IgA)
Description: Antirotavirus immunoglobulin A (IgA) and IgG were measured by enzyme-linked immunosorbent assay at the Laboratory of Specialized Clinical Studies at the Cincinnati Children's Hospital Medical Center (Cincinnati, Ohio). A standard serum pool was used to determine arbitrary units of rotavirus IgA or IgG in each sample. A subject was considered seropositive if the IgA or IgG rotavirus antibody concentration was ≥20 U/mL.
Time Frame: Visit 1 (pre-vaccination) and 8 weeks post vaccination
Population: All participants meeting inclusion/exclusion criteria and with valid samples.
Measure: Count of Participants; unit: Participants
Groups:
- Measles-rubella and Rotavirus Vaccine: receive one 0.5 ml subcutaneous dose of live attenuated measles-rubella vaccine and one 1.0 ml dose of oral Rotarix vaccine at 9 months of age
  Rotarix vaccine: one 1.0 ml dose of oral rotavirus vaccine at 9 months of age
  measles-rubella vaccine: one 0.5 ml subcutaneous dose of live attenuated measles-rubella vaccine
Arm/Group | Measles-rubella and Rotavirus Vaccine | Measles-rubella Vaccine
Number analyzed (Participants) | 239 | 240
Participants
  Pre-vaccination: Seropositive | 126 | 113
  Pre-vaccination: Not seropositive | 113 | 127
  Post-vaccination: number analyzed (Participants) | 230 | 240
  Post-vaccination: Seropositive | 160 | 110
  Post-vaccination: Not seropositive | 70 | 130

6. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-rotavirus Immunoglobulin A (IgA)
Description: Antirotavirus immunoglobulin A (IgA) and IgG were measured by enzyme-linked immunosorbent assay at the Laboratory of Specialized Clinical Studies at the Cincinnati Children's Hospital Medical Center (Cincinnati, Ohio). A standard serum pool was used to determine arbitrary units of rotavirus IgA or IgG in each sample. Rotavirus IgA and IgG values of <20 U/mL are converted to 10 U/mL for calculation purposes.
Time Frame: Visit 1 (pre-vaccination) and 8 weeks post vaccination
Population: All participants meeting inclusion/exclusion criteria and with valid samples.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 239 | 240
U/mL
  Pre-vaccination | 43.6 [34.8 to 54.5] | 39.2 [31.3 to 49.1]
  Post-vaccination | 60.6 [49.4 to 74.2] | 38.1 [30.5 to 47.6]

7. Secondary Outcome: Percentage/Number of Subjects Seropositive for Anti-rotavirus Immunoglobulin G (IgG)
Description: as for outcome 5
Time Frame: Visit 1 (pre-vaccination) and 8 weeks post vaccination
Population: All participants meeting inclusion/exclusion criteria and with valid samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 240 | 240
Participants
  Pre-vaccination: Seropositive | 159 | 140
  Pre-vaccination: Not seropositive | 81 | 100
  Post-vaccination: number analyzed (Participants) | 231 | 236
  Post-vaccination: Seropositive | 204 | 135
  Post-vaccination: Not seropositive | 27 | 101

8. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-rotavirus Immunoglobulin G (IgG)
Description: as for outcome 6
Time Frame: Visit 1 (pre-vaccination) and 8 weeks post vaccination
Population: All participants meeting inclusion/exclusion criteria and with valid samples.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 240 | 240
U/mL
  Pre-vaccination | 79.2 [61.4 to 102.1] | 63.2 [49.1 to 81.4]
  Post-vaccination | 168.6 [137.3 to 207.2] | 60.1 [46.7 to 77.5]

9. Secondary Outcome: Percentage/Number of Subjects With Seroconversion for Anti-rotavirus Immunoglobulin A (IgA)
Description: as for outcome 5
Time Frame: 8 weeks post vaccination
Population: All subjects that met inclusion and exclusion criteria with valid samples and were not seropositive prior to the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 110 | 126
Participants
  Seroconversion | 48 | 8
  No seroconversion | 62 | 118

10. Secondary Outcome: Percentage/Number of Subjects With Seroconversion for Anti-rotavirus Immunoglobulin G (IgG)
Description: as for outcome 5
Time Frame: 8 weeks post vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 80 | 99
Participants
  Seroconversion | 55 | 7
  No seroconversion | 25 | 92

11. Secondary Outcome: Number/Percentage of Subjects Experiencing Immediate Post-vaccination Reactions Following Administration of Vaccine
Description: Immediate reactogenicity was defined as local or systemic reactions occurring directly and up to 30 minutes after vaccine receipt, with an emphasis on allergic reactions.
Time Frame: 30 minutes post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 240 | 240
Participants
  Any immediate reaction | 0 | 0
  No immediate reaction | 240 | 240

12. Secondary Outcome: Number/Percentage of Subjects Experiencing Solicited Adverse Events
Description: Solicited non-serious adverse events were collected based on recall at study visits 2 (Day 4) through 5 (Day 14) following administration of Rotarix® vaccine. They included diarrhea, fever, vomiting, loss of appetite, irritability, and intussusception. Adverse events were graded for severity and relationship to vaccine.
Time Frame: 14 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 240 | 240
Participants
  Grade 1: unrelated to vaccine | 25 | 34
  Grade 2: unrelated to vaccine | 4 | 4
  Grade 3: unrelated to vaccine | 2 | 0
  None | 209 | 202

13. Secondary Outcome: Number/Percentage of Subjects Experiencing Unsolicited Non-serious Adverse Events
Description: Solicited non-serious adverse events were collected based on recall at study visits 2 (Day 4) through 5 (Day 14) following administration of Rotarix® vaccine. Adverse events were graded for severity and relationship to vaccine.
Time Frame: 14 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 240 | 240
Participants
  Related to vaccine | 0 | 0
  Unrelated to vaccine | 63 | 68
  No unsolicited non-serious adverse event | 177 | 172

14. Secondary Outcome: Number/Percentage of Subjects Experiencing Serious Adverse Events
Description: An adverse event (AE) or suspected AE was considered "serious" if it resulted in any of the following outcomes:
  * Death
  * A life-threatening AE (the term "life-threatening" in the definition of "serious" refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  Important medical events that may not result in death, be life threatening, or require hospitalization would have been considered severe adverse events when, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: 2 months after vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 240 | 240
Participants
  Any serious adverse event, unrelated to vaccine | 10 | 6
  No serious adverse event | 230 | 234

15. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Measles Virus Serum Neutralization Antibodies
Description: Sera were analyzed for the presence of measles virus serum neutralizing antibodies (SNAs), using a standardized plaque reduction neutralization (PRN) assay, in which PRN titers, defined as the serum dilutions that reduced the number of plaques by 50%, were calculated using the Kärber method [12]. A 1:100 dilution of World Health Organization (WHO) Second International Standard Anti-Measles Serum (IS, coded 66/202, supplied by the National Institute for Biological Standards and Control, South Mimms, United Kingdom) was tested in parallel with each serum specimen to calculate the reciprocal of the 50% end point titer determined by the PRN test.
Time Frame: 8 weeks post vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
Number analyzed (Participants) | 227 | 233
mIU/mL | 196.3 [175.3 to 219.7] | 194.2 [174.0 to 216.7]

16. Other Pre Specified Outcome: Number of Participants With Rotavirus Vaccine Shedding
Description: Based on 5 grams of stool sample. Vaccine shedding defined as presence of vaccine-type rotavirus in stool at 4 (+/-1) and/or 7 (+/-1) days post rotavirus vaccination detected by enzyme-linked immunosorbent assay (ELISA) and typed by reverse-transcriptase polymerase chain reaction (RT-PCR).
Time Frame: Day 0, Day 4 and Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Measles-rubella and Rotavirus Vaccines
Number analyzed (Participants) | 240
Participants
  Day 0: Negative | 140
  Day 0: Positive | 0
  Day 0: No stool | 100
  Day 4: Negative | 234
  Day 4: Positive | 4
  Day 4: No stool | 2
  Day 7: Negative | 234
  Day 7: Positive | 6
  Day 7: No stool | 0

ADVERSE EVENTS:
Time Frame: 2 months after vaccination
Description: Local and systemic adverse events were assessed on days 4, 7, 11, 14, and 28 after vaccination through home visits by trained field workers. Solicited adverse events includes diarrhea, fever, vomiting, loss of appetite, irritability, and signs of intussusception (colicky abdominal pain or paroxysms of crying/screaming, abdominal distension or mass, intermittent irritability or lethargy with behavioral changes, stool with blood or "red currant jelly," and/or vomiting ≥2 episodes/day).
Arm/Group | Measles-rubella and Rotavirus Vaccines | Measles-rubella Vaccine
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/240
Serious Adverse Events (participants affected / at risk) | 10/240 | 6/240
Other Adverse Events (participants affected / at risk) | 63/240 | 68/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Measles-rubella and Rotavirus Vaccines (N=240) | Measles-rubella Vaccine (N=240)
Acute bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Acute nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute watery diarrhea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia with UTI (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Severe pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Measles-rubella and Rotavirus Vaccines (N=240) | Measles-rubella Vaccine (N=240)
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dysentery (Gastrointestinal disorders) | 9 | 12
Ear pain (Ear and labyrinth disorders) | 1 | 0
Fungal infection (Infections and infestations) | 2 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 32 | 38
Oral candidiasis (Gastrointestinal disorders) | 1 | 0
Otitis media chronic (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract infection (Infections and infestations) | 16 | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No